CLINICAL TRIAL: NCT04806958
Title: Evaluating the PulsePoint Mobile Device Application to Increase Bystander Resuscitation for Victims of Sudden Cardiac Arrest
Brief Title: The PulsePoint Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Steven Brooks (Other)
Collaborators: University of British Columbia (Other); BC Emergency Health Services (Unknown); Winnipeg Fire Paramedic Service (Unknown); University of Manitoba (Other); University of Toronto (Other); Ohio State University (Other); Columbus Division of Fire (Unknown); PulsePoint Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Steven Brooks, Associate Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 148168
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Heart Arrest; Heart Diseases; Cardiovascular Diseases
Keywords: Cardiac Arrest; Cardiopulmonary Resuscitation; Automated External Defibrillators; Smartphones
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, EMS providers, dispatch providers, treating physicians will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Emergency Dispatch PLUS PulsePoint notification (Experimental): Eligible 911 calls randomized to the experimental arm of the study will undergo usual dispatch of emergency services personnel as per pre-existing local protocols and activation of the PulsePoint system. When triggered, the system will push location data to all PulsePoint mobile application users within 400 meters of the emergency. Devices receiving the alerts from the PulsePoint system will alarm with auditory, tactile and visual stimuli. The application will present a map showing the exact location of the emergency and the closest public access defibrillator.
  Interventions: Other: PulsePoint notification
- Conventional Emergency Dispatch (No Intervention): Patients randomized to the control arm will receive conventional emergency medical dispatching procedures as per pre-existing local protocols (e.g. dispatch of emergency vehicles, attempted dispatch-assisted CPR) without activation of the PulsePoint system. 911 calls randomized to the control arm will not be associated with any PulsePoint alerts.

INTERVENTIONS:
Other: PulsePoint notification — The PulsePoint interface software monitors each 9-1-1 call on dispatch computers and is automatically triggered by particular conditions including call type (e.g. suspected cardiac arrest) and location type (public location). When triggered, the system pushes location data to all PulsePoint mobile application users within 400 meters of the emergency location.
  When a mobile device running the PulsePoint Respond application receives the alert data from the PulsePoint system, the device alarms with auditory, tactile (vibration) and visual stimuli. The application presents a map showing the exact location of the suspected cardiac arrest and the closest public access defibrillator.
  Arms: Conventional Emergency Dispatch PLUS PulsePoint notification

SUMMARY:
This randomized controlled trial will evaluate whether use of the PulsePoint system increases bystander CPR or defibrillator use compared to standard dispatch procedures in patients who suffer non-traumatic, out-of-hospital cardiac arrest in a public location. Half of all suspected cardiac arrest 9-1-1 calls in a public location will receive PulsePoint alerts (treatment arm). The other half of this eligible patient cohort will receive standard dispatch procedures (control arm).

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) is a major public health problem. More than 45,000 Canadians suffer OHCA annually, with only 8.4% surviving to hospital discharge. Early bystander cardiopulmonary resuscitation (CPR) and defibrillator use can save lives but are rarely done.

Advances in mobile device technology have allowed the development of a system which can notify CPR-trained citizens within 400 meters of a possible cardiac arrest. The PulsePoint mobile device application (www.pulsepoint.org) empowers them to respond and provide basic life support while professional crews are being dispatched. When a mobile device receives the alert data from the PulsePoint system, the application presents a map showing the exact location of the emergency and the closest public access defibrillator.

PulsePoint will be implemented in 2 regions across Canada and the US (British Columbia and Columbus, Ohio). After a coordinated marketing campaign in each participating region to maximize the number of mobile device application downloads in the community, 9-1-1 calls for suspected cardiac arrest will be randomized to conventional dispatch for suspected cardiac arrest versus conventional dispatch plus PulsePoint notifications. The primary outcome will be bystander CPR or defibrillator use prior to professional responders arriving on scene. The primary analysis will involve comparing outcomes between the control and treatment groups among randomized patients who satisfy inclusion and exclusion criteria and have at least one PulsePoint responder within 400 meters of the cardiac arrest event.

The investigators hypothesize that the PulsePoint system will have an immediate impact on increasing bystander CPR and defibrillator use in participating communities. In the long term, this project will provide valuable data on how effective PulsePoint is with respect to bystander resuscitation and survival. The data will directly inform policy decisions about PulsePoint implementation in the participating communities and guide other North American jurisdictions around these policy decisions in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with 911 calls assigned as "suspected" or "confirmed" cardiac arrest and,
2. Are confirmed to be EMS-treated, public location out-of-hospital cardiac arrest.

Exclusion Criteria:

1. Traumatic cardiac arrest, or
2. Cardiac arrests occurring in the context of a dangerous scene as determined by the 9-1-1 call-taker, or
3. EMS-witnessed cardiac arrest, or
4. Cardiac arrests not treated by EMS ("Do Not Resuscitate", signs of obvious death), or
5. Cardiac arrests occurring in nursing homes and health care facilities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving bystander resuscitation | Patients will be followed for this outcome during the interval from 9-1-1 call to emergency medical services arrival, an expected average of 5 minutes.
  Defined as the occurrence of either bystander CPR (chest compressions and or ventilations) or bystander application of a defibrillator prior to the arrival of emergency medical services.

SECONDARY OUTCOMES:
Proportion of patients receiving bystander CPR (secondary effectiveness outcome) | Patients will be followed for this outcome during the interval from 9-1-1 call to emergency medical services arrival, an expected average of 5 minutes.
  Defined as the occurrence of bystander CPR (chest compressions and or ventilations) prior to the arrival of emergency medical services.
Proportion of patients receiving bystander defibrillator use (secondary effectiveness outcome) | Patients will be followed for this outcome during the interval from 9-1-1 call to emergency medical services arrival, an expected average of 5 minutes.
  Defined as bystander application of defibrillator pads on the chest of the victim prior to the arrival of emergency medical services.
Proportion of patients receiving bystander defibrillator shock delivered (secondary effectiveness outcome) | Patients will be followed for this outcome during the interval from 9-1-1 call to emergency medical services arrival, an expected average of 5 minutes.
  Defined as the occurrence of a bystander applying an automated external defibrillator and then applying a defibrillatory shock to the chest of the victim.
Proportion of patients with return of spontaneous circulation (secondary effectiveness outcome) | Patients are followed from EMS arrival on scene until arrival at hospital, an expected average of 35 minutes.
  Defined as any palpable pulse or measurable blood pressure.
Proportion of patients surviving to hospital discharge (secondary effectiveness outcome) | Patients are followed until death or discharge from hospital, an expected average of 30 days.
  Defined as survival of a patient to the point of discharge from the acute care hospital. Discharge may be to a residence or long term care facility.
Proportion of patients surviving to hospital discharge with good functional outcome (secondary effectiveness outcome) | Patients are followed until death or discharge from hospital, an expected average of 30 days.
  Defined as the occurrence of a patient surviving to hospital discharge with a Cerebral Performance Score of 1 or 2.
EMS response time interval (secondary safety outcome) | Expected average of 5 minutes.
  Defined as the time interval between the 9-1-1 call and the EMS arrival on scene.
EMS on scene time interval (secondary safety outcome) | Expected average of 30 minutes.
  Defined as the time interval between the EMS arrival on scene to EMS departure from scene.
Proportion of patients receiving bystander interference with the resuscitation effort (secondary safety outcome) | Patients will be followed for this outcome in the time interval between 9-1-1 call and EMS departure from scene, an expected average of 35 minutes.
  Defined as emergency medical service crew reports of bystander interference with the resuscitation effort.
Number of PulsePoint application downloads (secondary system performance outcomes) | Downloads in the participating communities will be tracked for the duration of the anticipated 2 year patient recruitment time frame.
  Defined as the number of PulsePoint application downloads in each participating community.
Number of PulsePoint application users notified (secondary system performance outcome) | This will be tracked for each notification event that occurs during the anticipated 2 year accrual time frame.
  The number of application users notified for each PulsePoint notification.
Sensitivity of PulsePoint activation (secondary system performance outcome) | This will be tracked for each notification event that occurs during the anticipated 2 year accrual time frame.
  The sensitivity of the PulsePoint activation as it relates to activation for true cardiac arrests.
False positive rate for PulsePoint activation (secondary system performance outcome) | This will be tracked for each notification event that occurs during the anticipated 2 year accrual time frame.
  The false positive rate for PulsePoint activation resulting from activation of the system for conditions other than cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Brooks, MD MHSc, Principal Investigator — Queen's University; John M Tallon, MD MSc, Principal Investigator — University of British Columbia
Locations (3):
- Columbus Division of Fire, Columbus, Ohio, United States
- Canada (2):
  - British Columbia Emergency Health Services, Vancouver, British Columbia
  - Winnipeg Fire Paramedic Service, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No